CLINICAL TRIAL: NCT03177278
Title: A Phase 1, Open-Label Study to Assess the Metabolism, Excretion, and Mass Balance of [14C]-Plazomicin Following a Single IV Infusion in Healthy Adult Male Subjects
Brief Title: A Study to Assess the Metabolism, Excretion, and Mass Balance of Radio-Labeled Plazomicin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACHN-490-010
Record Dates: First submitted 2017-06-01; First posted 2017-06-06 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: [14C]-plazomicin

INTERVENTIONS:
Drug: [14C]-plazomicin — single intravenous dose

SUMMARY:
This is a single-center, open label, non-randomized metabolism, excretion, and mass balance study of a single IV infusion of [14C]-plazomicin in healthy, adult male subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Medically healthy, with no clinically significant medical history, physical examination findings, vital signs or ECG findings

Key Exclusion Criteria:

* Use of tobacco- or nicotine-containing products
* Has received radio-labeled substances or has been exposed to radiation sources within 12 months of dosing or is likely to receive radiation exposure or radioisotopes within 12 months of dosing such that participation in this study would increase their total exposure beyond the recommended levels considered safe
* History of hearing loss or a family history of hearing loss, or a prior diagnosis of sensorineural hearing loss or Ménière's disease
* History in the past 90 days of prior trauma to the outer or internal structures of the ear or tinnitus
* History or family history of vestibular disorder, chronic vertigo (sensation of spinning), chronic dizziness

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Due to nature of radio-labeled drug studies and the inherent risk to fertility and reproduction, females are ineligible to participate in this study
Enrollment: 6 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Sum of percent of total radioactivity recovered in urine and feces relative to the administered radioactive dose minus any radioactivity lost due to emesis | 15 days
Total radioactivity concentration equivalents in plasma and blood | 15 days
Plazomicin concentrations in plasma and urine | 15 days

SECONDARY OUTCOMES:
Incidence and severity of adverse events | 21 days
Change from baseline in vital signs post dose (temperature, pulse, respiration, blood pressure) | 1 day
Absolute values of and change from baseline in clinical laboratory values (hematology, serum chemistry, urine analysis) | 4 days
Physical examination | Screening

CONTACTS AND LOCATIONS:
Overall Officials: Shyeilla Dhuria, Study Director — Achaogen, Inc.
Locations (1):
- Clinical Site, Lincoln, Nebraska, United States